CLINICAL TRIAL: NCT06630949
Title: Using a Novel Method to Diagnose the Prevalence and Health Impact of Muscle Loss in Older Adults
Brief Title: D3-Creatine and Skeletal Muscle in Older Adults
Acronym: D3-Cr
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor and Canada Research Chair, McMaster University
Other Study IDs: 14733
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Aging; Muscle Loss
Keywords: aging; muscle; stable isotope tracer; mobility; sarcopenia; creatine; creatinine
MeSH Terms: conditions — Muscular Atrophy; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and bloodspot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The age-related decline in muscle mass and strength are collectively referred to as sarcopenia. However, the tools currently employed to assess skeletal muscle mass (SMM) (e.g., Dual-energy Xray Absorptiometry; DXA) have substantial drawbacks, and it is known that DXA-lean soft tissue (LST) is generally not associated with health outcomes of interest. Thus, the investigators propose using a novel, non-invasive, stable isotope-labelled probe (Deuterium (D)-labelled creatine (D3-creatine; D3-Cr)) to measure skeletal muscle mass in a large cohort of older individuals. The development and employment of new methods to accurately quantify the biological substrate of sarcopenia, skeletal muscle, are critical for the measure to remain clinically relevant. The plan is to measure 350 persons from the recently established (M3) prospective cohort. There will be measurement of lean soft tissue LST and appendicular LST (aLST) using DXA and compared to D3-Cr-measured SMM (D3-Cr-SMM) at baseline, 12mo, and 24mo (2yr) of follow-up. Physical mobility will also be measured (using various instruments).

DETAILED DESCRIPTION:
The tools currently employed to assess skeletal muscle mass (SMM), including DXA, have substantial drawbacks. DXA does not measure muscle per se but provides an assessment of lean soft tissue (LST) as a proxy for skeletal muscle. Even if confined to the appendages (aLST), DXA assessments include many non-muscle constituents (e.g., connective tissue, water), which are poorly and inconsistently related to mobility and falls with aging. As a superior measure to DXA, the investigators will use a novel, stable isotope-labelled probe to measure SMM. This method uses the oral ingestion of a small dose of deuterium (D)-labelled creatine (D3-creatine; D3-Cr), which is irreversibly converted to creatinine when taken up by skeletal muscle. The dilution of the labelled creatinine provides a safe, non-invasive, and highly accurate measure of SMM. The utilization of D3-Cr-measured SMM (D3-Cr-SMM) requires no specific diet and requires only the collection of a spot urine sample.

The plan is to recruit a sub-sample of older Canadians between 60 and 80 living in the greater Hamilton-Toronto area. Participants will be recruited through the MacM3 (M3) cohort study. MacM3 will enroll a sample of 2,000 participants from a pre-recruited representative sample of more than 10,000 older adults living in the greater Hamilton and Toronto areas who consented to be contacted for further research as part of a larger research platform. From this pool of 2000 individuals in MacM3, the plan is to recruit 350 people. Participants will be classified across the three levels of mobility limitations based on the MacM3 screening criteria of preclinical mobility limitation (i.e., able to manage without difficulty - no mobility limitation, able to manage without difficulty but sometimes with task modification - early mobility limitation, and able to manage with minor difficulty - minor mobility limitation, which will provide valuable insight into whether changes in D3-Cr-SMM are associated with a change in categorical mobility status.

The proposed research design is a prospective cohort study including 350 older (65-80 y) men and women. All participants will undergo muscle mass assessments via D3-Cr, body composition (LST, aLST, fat mass) via DXA, and dietary intake by 24h recall (ASA24) at baseline, 1y and 2y of follow-up. Performance-based assessments of physical function, mobility status and muscular strength will also be conducted at baseline, 1y and 2y of follow-up. During the quarterly follow-up phone calls, all participants will be screened limitation screening questions (see inclusion criteria), allowing us to capture changes in mobility status (i.e., no, early, minor or major mobility limitation) over time.

ELIGIBILITY:
Inclusion Criteria:

Participants will be considered eligible for this study if they are

* Between 60 and 80y (inclusive),
* Reside in the local (i.e., within 60km of Hamilton) community; and
* Are willing and able to provide written informed consent.

Participants must fall into one of three self-reported mobility limitations based on validated screening criteria via a structured phone interview. Potential participants will be asked whether they have any difficulty:

* Walking 800m;
* Climbing ten steps; and
* Transferring from/into a car or bus.

Response options include:

* Managing without difficulty;
* Managing without difficulty but with task modification; or
* Managing with minor difficulty.

Exclusion Criteria:

* Participants who self-report more than minor difficulty will be considered to have a mobility disability and excluded.
* Participants who cannot speak or read English will also be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be a sub-sample from the McMaster Monitoring My Mobility (MacM3) cohort, a newly founded research cohort. The MacM3 cohort is a longitudinal study of community-dwelling older Canadians (age 60-80 y at baseline) with different levels of mobility limitation (i.e., able to manage without difficulty - no mobility limitation; able to manage without difficulty but with task modification - early mobility limitation; and able to manage with minor difficulty - minor mobility limitation) collecting detailed mobility and health data on participants over two years of follow-up.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 2 years
  D3-creatine-measured muscle mass
Lean tissue mass | 2 years
  DXA-measured lean tissue mass

SECONDARY OUTCOMES:
Questionnaire Mobility | 2 years
  Questionnaire-based assessment of participant's physical mobility
SPPB | 2 years
  Short physical performance battery (SPPB)
Timed up and go | 2 years
  Participant starts in a seated position, stands up upon go signal, walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Principal Investigator — McMaster University, Department of Kinesiology
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will evaluate all requests to obtain IPD when the study is complete.